CLINICAL TRIAL: NCT06539130
Title: Medical Practices and Representations of People From Haiti Living With or Without HIV or Chronic HBV
Brief Title: Medical Practices and Representations of People From Haiti in French Guiana
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Other Study IDs: Parcours Quali
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Social Representations of Infectious Diseases
Keywords: Migration; Infectious disease; Traditional medecine; Precariousness
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational, cross-sectional, qualitative study of the population of Haitian origin living in French Guiana and the professionals working with them

DETAILED DESCRIPTION:
French Guiana is an overseas department located in South America, in the heart of the Amazon, between Brazil and Suriname. In terms of surface area (83,846 km2), it is the second largest region in France, but also one of the least densely populated, with 290,691 inhabitants in January 2020.

The region has undergone several waves of migration, and almost 38% of its current population born abroad. It is estimated that more than 10% of the population is of Haitian origin in 2020, although these figures do not include the number of illegal immigrants. The first major waves of migration date back to the early 1980s, in connection with political unrest in Haiti. The last major wave of Haitian migration took place in 2015-2016, following the tightening of Dominican migration policy and the expulsion of more than 100,000 Haitian nationals to Haiti.

However, despite the importance of the demographic component of Haitian origin in the Guianese population as a whole, relatively few studies have focused on the care practices inherent in this cultural community. Despite the importance of care using plants in Haiti, particularly given the difficulties in accessing biomedical care, only a few and/or relatively old ethnobotanical works, for example, address the question of Haitian phytotherapy.

The glaring lack of recent work on Haitian ethnomedicine was therefore a trigger for initiating this qualitative study, as part of a more global approach to deciphering the life and care paths followed by people originally from Haiti ("Parcours d'Haïti" study, main protocol).

In addition, people from Haiti have high levels of HIV and hepatitis B virus infection. Yet the anthropology of health and social epidemiology have largely demonstrated the weight of economic, political, cultural and social determinants (such as gender, age, administrative status, housing, social support, activity and standard of living) - which make up what is called the "political space of health" - on social inequalities in health. These inequalities, whether gendered, generational, geographical or socio-cultural, have been highlighted in relation to the higher prevalence of HIV infection among people from sub-Saharan Africa living in France or people from Haiti living in the French West Indies.

A better understanding of the level of knowledge of these two diseases, their social and cultural representations, and the attitudes and behaviours relating to their prevention is necessary in order to adapt prevention and health communication strategies. Few studies have explored these areas of knowledge.

Health, social work and voluntary sector professionals involved in providing medico-psychosocial support to people from Haiti report difficulties of a cultural nature and relating to health literacy, although these representations and their impact on practice have not been studied further.

ELIGIBILITY:
People originated from Haïti Inclusion Criteria:

* To be born in Haïti
* To have moved to French Guiana for more than 3 months
* To be more than 18 years old
* To be infected or not by HIV or HBV
* To agree to participate to the study

Health and social professionals Inclusion Criteria:

* To be a health or social professional
* To be involved in medico-psycho-social care to people originated from Haïti
* To be more than 18 years old
* To agree to participate to the study

Exclusion Criteria:

* Not to be able to answer the questoins in French or Haïtian creole langage
* To be under guardianship, curatorship or legal protection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People originated from Haïti Health and social professionals working with people originated from Haïti
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
Description of social representations of HIV and HBV infections among migrant population from Haïti | At inclusion
  To describe the social representations of HIV and HBV infections and their impact on use of traditional medecine among migrant population from Haïti, using qualitative questionnaire

SECONDARY OUTCOMES:
Description of living conditions of migrants from Haïti | At inclusion
  To describe living conditions and health seeking behavior of migrants from Haïti after their arrival in French Guiana using a qualitative questionnaire
Description of difficulties to access health care and health prevention | At inclusion
  To describe difficulties met by migrants from Haïti after their arrival in French Guiana to access health care and health prevention using a qualitative questionnaire
Description of food insecurity situations met by migrants from Haïti | At inclusion
  To describe food insecurity situations and coping strategies met by migrants from Haïti after their arrival in French Guiana using a qualitative quesitonnaire
Description of social and health professionals representations on migrants from Haïti | At inclusion
  To describe representations from health and social professionals working with migrants from Haïti usng a qualitative questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Adenis, MD, PhD, Study Director — Centre Hospitalier de Cayenne
Locations (1):
- Centre Hospitalier de Cayenne, Cayenne, French Guiana

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tareau MA, Greene A, Palisse M, Odonne G. Migrant Pharmacopoeias: An Ethnobotanical Survey of Four Caribbean Communities in Amazonia (French Guiana). Econ Bot. 2022;76(2):176-188. doi: 10.1007/s12231-021-09529-0. Epub 2021 Oct 20. PMID 34697504
- [Background] Weniger B, Rouzier M, Daguilh R, Henrys D, Henrys JH, Anton R. [Traditional medicine in the Central Plateau of Haiti. 2. Ethnopharmacologic inventory]. J Ethnopharmacol. 1986 Jul;17(1):13-30. doi: 10.1016/0378-8741(86)90070-x. French. PMID 3762193
- See also: Discriminations and access to health care in French Guiana — https://www.cairn.info/revue-cahiers-de-la-lcd-lutte-contre-les-discriminations-2017-3-page-174.htm
- See also: Urban medicinal gardens in French Giuana : an Haïtian network — https://core.ac.uk/download/pdf/15518775.pdf
- See also: Contemporary images of urban poverty in France, the United States and Latin America — https://www.ias.edu/sites/default/files/sss/pdfs/Fassin/Exclusion-underclass-marginalidad.pdf
- See also: HIV/AIDS at the Europe's caribbean borders. Memories of an epidemic in a land of exception — https://journals.openedition.org/anthropologiesante/7608
- See also: The migrant couple confronted with HIV — https://www.persee.fr/doc/homig_1142-852x_2006_num_1262_1_4494